CLINICAL TRIAL: NCT03962257
Title: Improving the Informed Consent Process for Infertile Patients Undergoing Assisted Reproductive Technology (ART) With EngagedMD
Brief Title: The Use of an Online Learning and Consent Platform in Infertility Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 18-3258
Record Dates: First submitted 2019-05-20; First posted 2019-05-24 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Patient Satisfaction
Keywords: Patient education
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing one group receiving standard care and the other with standard care with the addition of the online learning platform
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention): This group will have standard of care infertility counseling and consent processes.
- Engaged MD (Experimental): This group will have standard of care infertility counseling and access to online teaching modules and the ability to sign consents online.
  Interventions: Other: EngagedMD online learning platform

INTERVENTIONS:
Other: EngagedMD online learning platform — The EngagedMD online learning platform is a compilation of learning modules and questions designed to give patients at-home access to visual and audio aids in infertility treatment. It also gives patients the ability to read and sign consents from home.
  Arms: Engaged MD

SUMMARY:
The primary purpose of this study is to objectively assess if interactive multimedia tutorials (online videos) enhances patients' comprehensive understanding of assisted reproductive technology (ART) adding EngagedMD, an online library of interactive videos, compared to the traditional process of consent and one-on-one teaching using a 15 question evaluation. The secondary outcome will be to qualitatively assess patients' overall experience of the teaching process comparing the addition of the EngagedMD content to solely traditional teaching for infertility treatment.

DETAILED DESCRIPTION:
Participants: This will be a multi-center trial with each center planning on recruiting 100 couples. Half of the couples will be planning on undergoing ovulation induction with insemination (OI/IUI) and the other half in-vitro fertilization (IVF).

Procedures (methods): This is a multi-center prospective randomized controlled trial where couples undergoing OI/IUI or IVF will be randomized to receiving the current traditional standard of in-person treatment teaching by their physician and nursing team with standard paper consents or to the identical process of in-person teaching with the addition of unrestricted access to the EngagedMD online video resource platform with online consents.

Patient demographics, knowledge base, psychological impact of with the treatment, teaching and the consent process and overall satisfaction with the process as a whole will be assessed using surveys administered at three time points throughout the treatment process. A subset of patients that agree will be contacted after the completion of the treatment cycle for a live phone interview.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be 18-49 years of age undergoing fertility treatment
* Able to give Informed Consent

Exclusion Criteria:

* Patients who do not have adequate command of the English language to provide informed consent

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Patient understanding | Each participant will be followed for one treatment cycle, or approximately 2-4 weeks.
  Patient understanding of infertility diagnoses and treatment by use of a pre and post test. The test comprises of 15 multiple choice questions and the patients will receive a score of 0-15 and this will be compared as a paired continuous variable from the pre-test score to their post-test score as well as an un-paired continuous variable between the conventional group and the EngagedMD group for pre- and post-test scores as well as delta scores between the two.

SECONDARY OUTCOMES:
Patient satisfaction | Each participant will be followed for one treatment cycle, or approximately 2-4 weeks.
  Patient satisfaction with their infertility treatment and consent processes will be assessed using questionnaires using a 5 point Likert scale progressing from very unsatisfied to very satisfied across a number of questions. The 5 point Likert questions will be assigned a value of 1-5 (with 1 being very unsatisfied and 5 being very satisfied) and will be assessed as a sum of points from the individual questions and compared as continuous variables between the conventional arm and the EngagedMD arm. There is an additional question asking patients to rank their satisfaction on a scale of 1-10 (with 1 being not satisfied at all and 10 being extremely satisfied) which will be used independently as a measure of patient satisfaction overall.

CONTACTS AND LOCATIONS:
Overall Officials: Linnea R Goodman, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Fertility CARE: The IVF Center, Winter Park, Florida
  - Positive Steps Fertility, Madison, Mississippi
  - UNC Fertility, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernard AL, Barbour AK, Meernik C, Madeira JL, Lindheim SR, Goodman LR. The impact of an interactive multimedia educational platform on patient comprehension and anxiety during fertility treatment: a randomized controlled trial. F S Rep. 2022 May 22;3(3):214-222. doi: 10.1016/j.xfre.2022.05.006. eCollection 2022 Sep. PMID 36212557